CLINICAL TRIAL: NCT00745355
Title: A Prospective Study of Quality of Life in Patients With Bladder Cancer
Brief Title: Quality of Life in Patients With Bladder Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Albert Einstein College of Medicine (Other); Northwell Health (Other); Lenox Hill Hospital (Other); DeltaQuest Foundation, Inc. (Unknown); Lahey Hospital & Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 08-076
Record Dates: First submitted 2008-08-22; First posted 2008-09-03 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Bladder Cancer
Keywords: Quality of Life; Questionnaires; 08-076
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: new patients with bladder cancer and/or are scheduled for radical cystectomy and urinary diversion
  Interventions: Behavioral: Quality Of Life questionnaires

INTERVENTIONS:
Behavioral: Quality Of Life questionnaires — All patients who agree to participate will be interviewed using a baseline idiographic quality of life assessment prior to surgery and at approximately 6, 12, 18 and 24 months postoperatively. All patients will also be asked to respond to a questionnaire including all standard measures (closed-ended, multiple choice items) before surgery and at approximately 3, 6, 12, 18 and 24 months post-surgery.

SUMMARY:
The purpose of this study is to learn about the quality of life of people living with bladder cancer. We are interested in learning about how the treatments for bladder cancer affect people. We plan to use the findings from this study to help doctors provide better care and information to patients with bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* All patients (male and female) who are diagnosed with bladder cancer
* Patients must be scheduled for radical cystectomy and urinary diversion are and/or being evaluated for neo-adjuvant chemotherapy prior to a planned cystectomy.
* Participants must be able to speak English.
* Participants must be able to provide informed consent.
* Participants must be 18 years of age or older to enroll.
* Participant may be eligible for and may receive neoadjuvant or adjuvant chemotherapy.
* Participant may have had intravesicle chemotherapy or immunotherapy (BCG, Interferon).

Exclusion Criteria:

* Subjects may be excluded from the study based on the following criteria:
* Follow-up care not obtained at MSKCC.
* Metastatic disease at diagnosis.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible MSKCC patients.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2008-08; Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Prospectively characterize the impact of radical cystectomy and different urinary diversions on quality of life of bladder cancer patients. | conclusion of study

SECONDARY OUTCOMES:
Compare various standard and idiographic measures of QOL, to determine their relative contributions in accounting for variance in key outcome criteria and prediction of patient QOL at subsequent assessment points. | conclusion of study
Examine how patients react to more in-depth probing of the interview associated with idiographic assessment. | conclusion of study
Develop a predictive model of QOL after radical cystectomy & urinary diversion using the data from idiographic and standard QOL measures. This model can ultimately be used in office based practice to guide treatment planning with each patient. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Bochner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

DOCUMENTS (1):
  • Informed Consent Form (2014-09-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT00745355/ICF_000.pdf